CLINICAL TRIAL: NCT05775367
Title: Cochlear Implantation in Infants and Toddlers With Single-Sided Deafness
Brief Title: Cochlear Implants in Young Children With SSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0862
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Single Sided Deafness; Unilateral Deafness; Hearing Loss, Unilateral; Hearing Loss; Congenital Hearing Loss; Deafness One Ear
Keywords: cochlear implant; uhl; ssd; children; hearing loss; deafness
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss; Articulation Disorders; Deafness | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: The study group will receive a cochlear implant under the age of three and be tested at the age of five. Two control groups, both five years old, will be tested as well. The control groups will consist of children with typical hearing in both ears and children with single-sided deafness who have not received a cochlear implant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Study Group (Experimental): This group of children with single-sided deafness will receive a cochlear implant.
  Interventions: Device: Cochlear Implant
- Typical Hearing Control Group (THCG) (No Intervention): This group of five-year-old children will have typical hearing in both ears.
- Single-Sided Deafness Control Group (SSDCG) (No Intervention): This group of five-year-old children will have single-sided deafness and no cochlear implant.

INTERVENTIONS:
Device: Cochlear Implant — A cochlear implant is a surgically implanted device that provides access to sound in people cannot get enough access to sound for communication with traditional hearing aids.
  Other Names: MED-EL SYNCHRONY 2 Cochlear Implant
  Arms: Study Group

SUMMARY:
The goal of this clinical trial is to investigate the safety and effectiveness of cochlear implantation in infants and toddlers with single-sided deafness.

The main questions it aims to answer are:

* Are cochlear implants an effective treatment of single-sided deafness in infants and toddlers?
* Are cochlear implants a safe treatment for single-sided deafness in infants and toddlers?

Participants will receive a cochlear implant and be followed until they are five years old. During those five years, the investigators will program the device and monitor auditory development.

Children will be asked to:

* Undergo cochlear implantation
* Wear their cochlear implant processor whenever they are awake.
* Participate in traditional hearing tests
* Participate in traditional hearing testing
* Participate in localization testing
* Participate in hearing in noise testing
* Participate in word recognition testing
* Participate in speech, language, and educational evaluations

The researchers will compare results to children with typical hearing in both ears and children with single-sided deafness who have not received an implant to observe any differences between the groups.

DETAILED DESCRIPTION:
Cochlear implantation is an FDA-approved option for children with single-sided deafness (SSD) who are over the age of five years. It has been well established that early implantation is advantageous for children with bilateral hearing loss as it takes advantage of the narrow window of neural plasticity. Research has yet to show the ideal age for implantation in children with SSD but considering the known impacts of age at implantation and duration of deafness on cochlear implant (CI) outcomes, five years is likely a late age for implantation in a child with congenital SSD. The purpose of this prospective clinical trial is to evaluate the safety and effectiveness of cochlear implantation in infants and toddlers with SSD.

Twenty (20) infants and Toddlers with SSD who are under the age of three will receive a cochlear implant. They will be followed until they reach the age of five. A group of typically hearing five-year-olds (n=20) and a group of five-year-olds with congenital or early onset SSD who have not received a cochlear implant (n=20) will also be recruited. All three groups of five-year-olds will be tested on measures of hearing in quiet, localizing, and hearing in spatially separated noise for comparison. Scores from the study group and the SSD control group will be compared to evaluate effectiveness.

The study will also explore the potential effects of SSD and early implantation on language, sensory processing, executive function, fatigue, and cognition.

ELIGIBILITY:
To be eligible to participate in this trial as a study subject, an individual must meet all of the following criteria:

1. Provision of signed and dated parental permission form
2. Unilateral severe-to-profound sensorineural hearing loss, congenital or acquired prior to the age of 2 years, defined as:

   1. Unaided residual hearing thresholds that yield a 3 frequency pure tone average (PTA; average at 500, 1000, and 2000 Hz) of ≥70 dB hearing loss (HL) in the ear to be implanted
   2. Hearing thresholds in the contralateral ear of ≤20 dB HL (3 frequency PTA of 500, 1000, and 2000 Hz).

   i. Thresholds should be measured using inserts wherever possible, or in the sound field to record the better-hearing ear alone. Required thresholds will include 250, 500, 1000, 2000, and 4000 Hz for air conduction. All other octave frequencies should be attempted. Bone conduction thresholds should be obtained at 500, 1000, 2000, and 4000 Hz. Masking should be attempted where appropriate. As participants are very young and masking is difficult for this population, suspected shadow audiograms will be sufficient if objective testing has confirmed a severe-to-profound unilateral hearing loss. Testing should confirm a severe-to-profound hearing loss, defined as a 3-frequency PTA (500, 1000, and 2000) >70 dB HL in one ear and ≤20 dB HL in the contralateral ear. The Primary Investigator and Lead Diagnostic Audiologist must agree on this diagnosis for enrollment.
3. Insufficient functional access to sound with appropriately fit amplification and aural habilitation (based on best practices and standard of care) defined as:

   1. PEACH + parent questionnaire scores below the expected value for children who lack the requisite language to complete open-set word recognition testing or
   2. Recorded Multisyllabic Lexical Neighborhood Test (MLNT) scores ≤ 30% in the ear to be implanted for children with the requisite language to complete open-set word recognition testing.
4. Between 7 months and 2 years, 11 months of age at implantation
5. Normal cochlear nerve as evaluated by imaging, required imaging by MRI brain/Internal auditory canal (IAC) without contrast with heavily weighted T2 images. CT optional at the physician's discretion.
6. No malformation of the cochlea
7. No evidence of progressive hearing loss of the contralateral ear
8. Willing to/has undergone hearing aid trial as warranted based on achieving an aided speech intelligibility index (SII) of > .65 when fitted via Desired Sensation Level (DSL) methods.
9. Realistic parental expectations: a verbal acknowledgment of the potential benefits and risks, and postoperative variation in performance. For instance, cochlear implantation will not restore normal hearing
10. Willing to obtain recommended meningitis vaccinations per Centers for Disease Control (CDC) recommendations
11. Development and cognition within the normal range as measured by the Developmental Assessment of Young Children (DAYC-2).
12. Parental commitment to study parameters including being able and willing to participate in the evaluation schedule, involvement in prescribed therapy, and travel to the investigational site and study-related activities. Parents must be willing to encourage wearing implant during waking hours.

To participate as an SSD control subject, an individual must meet all the following criteria:

1. Provision of signed and dated parental permission form
2. Unilateral severe-to-profound hearing loss - congenital or acquired prior to 2 years of age.

   1. Unaided residual hearing thresholds that yield a 3 frequency PTA (500, 1000, and 2000 Hz) of ≥70 dB HL in the affected ear.
   2. Hearing thresholds in the contralateral ear of ≤20 dB HL (3 frequency PTA of 500, 1000, and 2000 Hz)
   3. Unable to use or benefit from traditional amplification
3. Five years of age at the time of testing
4. Development and cognition within the normal range as measured by the Early Stanford Binet 2 (SB2).

To participate as a TH control subject, an individual must meet all the following criteria:

1. Provision of signed and dated parental permission form
2. Bilateral hearing thresholds that yield a PTA of ≤20 dB HL (3 frequency PTA of 500, 1000, and 2000 Hz).
3. Five years of age at the time of testing
4. Development and cognition within the normal range as measured by the Early SB2.

An individual who meets any of the following criteria will be excluded from participation in this study as a study subject:

1. English is not primary language of the home

   1. Speech perception materials are presented in English
   2. Parental questionnaires are administered in English
2. Conductive hearing loss in either ear
3. Cochlear nerve deficiency
4. Ossification/Fibrosis of the cochlea precluding implantation
5. Inability to participate in follow-up procedures (i.e., unwillingness, geographic location)
6. History of refractory chronic otitis media or condition that contraindicates anesthesia

An individual who meets any of the following criteria will be excluded from participation in this study as a control subject:

1. English is not primary language of the home

   1. Speech perception materials are presented in English
   2. Parental questionnaires are administered in English
2. Inability to participate in testing (i.e., unwillingness)

Ages: 7 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Mean Difference in the Signal-to-Noise Ratio 50 (SNR-50) between the Study Group and SSD Control Group as Measured with the BKB-SIN at 5 Years of Age | 5 years of age
  Two ½ lists of the Bamford-Kowal-Bench Speech in Noise Test (BKB-SIN) will be presented in a single condition: speech in front and masker directed 90 degrees to the normal ear. The SNR-50 represents the signal-to-noise ratio required to perceive 50% of the sentence. A lower score is better. All participants will be 5 years old at the time of testing. The study group will use their cochlear implant in conjunction with the normal hearing ear. The SSD control group will use their normal hearing ear alone.
Mean Difference in Localization Error Between the Study Group and the SSD Control group Measured at 5 Years of Age | 5 years of age
  Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 70 decibel (dB) sound pressure level (SPL) in a sound treated room. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. All participants will be 5 years old at the time of testing. The study group will use their cochlear implant in conjunction with the normal hearing ear. The SSD control group will use their normal hearing ear alone.

SECONDARY OUTCOMES:
Proportion of Procedural Related Adverse Events 6 months after Surgery | 6 months after surgery
  Procedural adverse events will be collected and reported as the proportion of subjects experiencing them.
Proportion of Device-Related Adverse Events 6 Months after Surgery | 6 months after surgery
  Device related adverse events will be collected and reported as the proportion of subjects experiencing them.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Park, AuD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The Children's Cochlear Implant Center at UNC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified raw data will be archived at Open Science Framework
Time Frame: At the time of the first publication following study closure
URL: https://osf.io/

REFERENCES:
- [Background] Bess FH, Tharpe AM. An introduction to unilateral sensorineural hearing loss in children. Ear Hear. 1986 Feb;7(1):3-13. doi: 10.1097/00003446-198602000-00003. PMID 3512353
- [Background] Bess FH, Tharpe AM. Unilateral hearing impairment in children. Pediatrics. 1984 Aug;74(2):206-16. PMID 6462820
- [Background] Corbin NE, Buss E, Leibold LJ. Spatial Hearing and Functional Auditory Skills in Children With Unilateral Hearing Loss. J Speech Lang Hear Res. 2021 Nov 8;64(11):4495-4512. doi: 10.1044/2021_JSLHR-20-00081. Epub 2021 Oct 5. PMID 34609204
- [Background] Anne S, Lieu JEC, Cohen MS. Speech and Language Consequences of Unilateral Hearing Loss: A Systematic Review. Otolaryngol Head Neck Surg. 2017 Oct;157(4):572-579. doi: 10.1177/0194599817726326. Epub 2017 Aug 22. PMID 28828919
- [Background] Lieu JEC. Permanent Unilateral Hearing Loss (UHL) and Childhood Development. Curr Otorhinolaryngol Rep. 2018;6(1):74-81. doi: 10.1007/s40136-018-0185-5. Epub 2018 Feb 15. PMID 29651362
- [Background] Purcell PL, Shinn JR, Davis GE, Sie KC. Children with unilateral hearing loss may have lower intelligence quotient scores: A meta-analysis. Laryngoscope. 2016 Mar;126(3):746-54. doi: 10.1002/lary.25524. Epub 2015 Oct 9. PMID 26452077
- [Background] Bell R, Mouzourakis M, Wise SR. Impact of unilateral hearing loss in early development. Curr Opin Otolaryngol Head Neck Surg. 2022 Oct 1;30(5):344-350. doi: 10.1097/MOO.0000000000000848. Epub 2022 Aug 24. PMID 36004776
- [Background] Russo FY, De Seta D, Orlando MP, Ralli M, Cammeresi MG, Greco A, de Vincentiis M, Ruoppolo G, Mancini P, Turchetta R. Hearing attention and quality of listening in children with unilateral hearing loss with and without hearing aid. Acta Otorhinolaryngol Ital. 2022 Apr;42(2):169-175. doi: 10.14639/0392-100X-N1746. PMID 35612509
- [Background] McKay S, Gravel JS, Tharpe AM. Amplification considerations for children with minimal or mild bilateral hearing loss and unilateral hearing loss. Trends Amplif. 2008 Mar;12(1):43-54. doi: 10.1177/1084713807313570. PMID 18270178
- [Background] Ead B, Hale S, DeAlwis D, Lieu JE. Pilot study of cognition in children with unilateral hearing loss. Int J Pediatr Otorhinolaryngol. 2013 Nov;77(11):1856-60. doi: 10.1016/j.ijporl.2013.08.028. Epub 2013 Sep 6. PMID 24035639
- [Background] Park LR, Griffin AM, Sladen DP, Neumann S, Young NM. American Cochlear Implant Alliance Task Force Guidelines for Clinical Assessment and Management of Cochlear Implantation in Children With Single-Sided Deafness. Ear Hear. 2022 Mar/Apr;43(2):255-267. doi: 10.1097/AUD.0000000000001204. PMID 35213890
- [Background] Brown KD, Dillon MT, Park LR. Benefits of Cochlear Implantation in Childhood Unilateral Hearing Loss (CUHL Trial). Laryngoscope. 2022 Mar;132 Suppl 6(Suppl 6):S1-S18. doi: 10.1002/lary.29853. Epub 2021 Sep 20. PMID 34542181
- [Background] Park LR, Dillon MT, Buss E, O'Connell BP, Brown KD. Spatial Release From Masking in Pediatric Cochlear Implant Recipients With Single-Sided Deafness. Am J Audiol. 2021 Jun 14;30(2):443-451. doi: 10.1044/2020_AJA-20-00119. Epub 2021 Mar 26. PMID 33769866
- [Background] Park LR, Preston E, Noxon AS, Dillon MT. Comparison of test methods to assess the implanted ear alone for pediatric cochlear implant recipients with single-sided deafness. Cochlear Implants Int. 2021 Sep;22(5):283-290. doi: 10.1080/14670100.2021.1903715. Epub 2021 Mar 24. PMID 33761831
- [Background] Nassrallah F, Tang K, Whittingham J, Sun H, Fitzpatrick EM. Auditory, Social, and Behavioral Skills of Children With Unilateral/Mild Hearing Loss. J Deaf Stud Deaf Educ. 2020 Apr 5;25(2):167-177. doi: 10.1093/deafed/enz041. PMID 31836889
- [Background] Bess FH, Davis H, Camarata S, Hornsby BWY. Listening-Related Fatigue in Children With Unilateral Hearing Loss. Lang Speech Hear Serv Sch. 2020 Jan 8;51(1):84-97. doi: 10.1044/2019_LSHSS-OCHL-19-0017. Epub 2020 Jan 8. PMID 31913803
- [Background] Hoff S, Ryan M, Thomas D, Tournis E, Kenny H, Hajduk J, Young NM. Safety and Effectiveness of Cochlear Implantation of Young Children, Including Those With Complicating Conditions. Otol Neurotol. 2019 Apr;40(4):454-463. doi: 10.1097/MAO.0000000000002156. PMID 30870355
- [Background] Deep NL, Purcell PL, Gordon KA, Papsin BC, Roland JT Jr, Waltzman SB. Cochlear Implantation in Infants: Evidence of Safety. Trends Hear. 2021 Jan-Dec;25:23312165211014695. doi: 10.1177/23312165211014695. PMID 34028328
- [Background] Chweya CM, May MM, DeJong MD, Baas BS, Lohse CM, Driscoll CLW, Carlson ML. Language and Audiological Outcomes Among Infants Implanted Before 9 and 12 Months of Age Versus Older Children: A Continuum of Benefit Associated With Cochlear Implantation at Successively Younger Ages. Otol Neurotol. 2021 Jun 1;42(5):686-693. doi: 10.1097/MAO.0000000000003011. PMID 33710159
- [Background] Benchetrit L, Ronner EA, Anne S, Cohen MS. Cochlear Implantation in Children With Single-Sided Deafness: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2021 Jan 1;147(1):58-69. doi: 10.1001/jamaoto.2020.3852. PMID 33151295